CLINICAL TRIAL: NCT00593814
Title: A Clinical Evaluation of the GORE EXCLUDER® Bifurcated Endoprosthesis - Low Permeability in the Primary Treatment of Infrarenal Abdominal Aortic Aneurysms
Brief Title: GORE EXCLUDER® Endoprosthesis - Low Permeability in Treatment of Abdominal Aortic Aneurysms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Lanesha Hill, WL Gore & Associates
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAA 04-04
Record Dates: First submitted 2007-12-20; First posted 2008-01-15 (Estimated); Results first posted 2010-08-23 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2017-12

CONDITIONS: Aortic Aneurysm, Abdominal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: GORE EXCLUDER® Bifurcated Endoprosthesis-Low Permeability — Implant

SUMMARY:
The purpose of this study is to evaluate the performance of the GORE EXCLUDER® Bifurcated Endoprosthesis-Low Permeability in the primary treatment of infrarenal abdominal aortic aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Infrarenal Abdominal Aortic Aneurysms less than 4.5 cm in diameter
2. Anatomy meets EXCLUDER Bifurcated Endoprosthesis - Low Permeability specification criteria per Instructions for Use
3. Access vessel able to receive 18 French introducer sheath
4. Life expectancy > 2 years
5. Appropriate candidate for endovascular repair
6. Ability to comply with protocol requirements including follow-up
7. 21 years of age or older, male or infertile female**

Exclusion Criteria:

1. Mycotic or ruptured aneurysm
2. Participating in another investigational device or drug study within one year
3. Documented history of drug abuse within six months
4. Myocardial infarction or cerebral vascular accident within six weeks
5. Pulmonary insufficiency requiring chronic home oxygen or inability to ambulate due to pulmonary function
6. Iliac anatomy that would require occlusion of both internal iliac arteries
7. Planned occlusion or reimplantation of significant mesenteric or renal arteries
8. Planned concomitant surgical procedure or previous major surgery within 30 days
9. Previous prosthesis placement in the aorta or iliac arteries
10. Degenerative connective tissue disease (e.g., Marfan's and Ehlers Danlos Syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2005-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark F Fillinger, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center

RESULTS

PARTICIPANT FLOW:
Groups:
- EXCLUDER Low Permeability: Modified EXCLUDER device with Low Permeability Layer designed to treat abdominal aortic aneurysms with an endovascular surgical technique. This device functions identically to the original EXCLUDER device, however, a low permeability film is included in the device to eliminate migration of serous fluid through the graft.
- Original EXCLUDER: Historical Sample from original study of EXCLUDER Device. The original EXCLUDER Device was designed for the endovascular treatment of abdominal aortic aneurysms.
Period: Overall Study
Arm/Group | EXCLUDER Low Permeability | Original EXCLUDER
Started | 139 | 120
Completed | 115 | 120
Not Completed | 24 | 0
Not completed — Death | 7 | 0
Not completed — Withdrawal by Subject | 7 | 0
Not completed — Lost to Follow-up | 7 | 0
Not completed — Physician Decision | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EXCLUDER Low Permeability | Original EXCLUDER | Total
Number analyzed (Participants) | 139 | 120 | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.9 (7.5) | 72.6 (7.7) | 73.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 14 | 41
  Male | 112 | 106 | 218
Region of Enrollment [Number; unit: participants]
  United States | 139 | 120 | 259

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Aneurysm Volume Increase Greater Than 10% at 2 Years Post-procedure
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | EXCLUDER Low Permeability | Original EXCLUDER
Number analyzed (Participants) | 104 | 102
participants | 9 | 31
Statistical Analysis 1: Comparison: EXCLUDER Low Permeability vs Original EXCLUDER; Test type: Superiority or Other; p < 0.001, Chi-squared

2. Secondary Outcome: Number of Subjects With Device Efficacy Events
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | EXCLUDER Low Permeability | Original EXCLUDER
Number analyzed (Participants) | 139 | 120
Participants | 14 | 19

ADVERSE EVENTS:
Arm/Group | EXCLUDER Low Permeability | Original EXCLUDER
Serious Adverse Events (participants affected / at risk) | 0/139 | 0/120
Other Adverse Events (participants affected / at risk) | 85/139 | 56/120
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EXCLUDER Low Permeability (N=139) | Original EXCLUDER (N=120)
Endoleak (Injury, poisoning and procedural complications) | 80 | 41
Increase in Aneurysm Diameter (Vascular disorders) | 2 | 24
Other (Social circumstances) | 7 | 0
Unplanned Branch Vessel Occlusion (Surgical and medical procedures) | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No